CLINICAL TRIAL: NCT06289465
Title: Investigation of the Effect of Working Style on Pain, Posture, Physical and Mental Status in Seasonal Hazelnut Workers
Brief Title: Examination of Pain, Posture, Physical and Mental Status in Seasonal Hazelnut Workers
Status: Completed | Type: Observational
Sponsor: Istanbul Bilgi University (Other)
Responsible Party: Principal Investigator, Furkan Çakır, Principal Investigator, Istanbul Bilgi University
Other Study IDs: IstanbulBU
Record Dates: First submitted 2024-02-25; First posted 2024-03-01 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-12

CONDITIONS: Agricultural Workers' Diseases; Posture; Pain; Depression; Fatigue
Keywords: agricultural workers; posture; pain; depression; fatigue
MeSH Terms: conditions — Agricultural Workers' Diseases; Pain; Depression; Fatigue | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Seasonal Workers (Experimental group): Criteria:
  * Volunteering to participate in the study.
  * To be between the ages of 18-34.
  * Having worked as a seasonal worker in Giresun for at least 1 month during the hazelnut harvest period.
  Interventions: Other: Observation
- Controls (Control group): Criteria:
  * Volunteering to participate in the study.
  * To be between the ages of 18-34.
  * Not having worked in any agricultural work during the summer period.
  * Living in the same socioeconomic environment as the group working as seasonal workers
  Interventions: Other: Observation

INTERVENTIONS:
Other: Observation — Seasonal workers will be assessed in the assessment area established in the hazelnut field and healthy controls will be assessed in their homes.

SUMMARY:
The collection of hazelnuts grown in our country provides a great source of employment for local people and seasonal workers. However, geographical conditions in hazelnut growing areas, challenging variable weather conditions in August and insufficient number of workers create a disadvantageous environment for seasonal workers.

In this study, it was aimed to investigate the effects of working conditions on mental status, fatigue, pain severity and postures (posture disorders, developmental delays, etc.) of young adults working in Giresun during the hazelnut picking season in comparison with the group living in the same sociodemographic and cultural environment but not working as seasonal workers.

DETAILED DESCRIPTION:
Agricultural work is a very broad concept that includes crop production as well as animal husbandry, forestry and aquaculture. An agricultural worker is a person who is unable to farm on his/her own account and tries to make a living by working for wages. A seasonal agricultural worker, on the other hand, is a person who works seasonally in someone else's agricultural field at any stage of agricultural production such as planting, cultivation, spraying, harvesting, in return for wages/wages or in-kind payment, permanently or on a mobile basis (Dedeoğlu & Bayraktar, 2019). The common point of seasonal agricultural workers, whether mobile or temporary, is that they cannot earn sufficient income from their own agricultural enterprises, they are families with little or no land, and they migrate seasonally (mobile) and/or temporarily (daily) to regions with more agricultural work opportunities in order to make a living.

Seasonal (mobile) agricultural workers usually stay in the places where they go to work until the work is finished. Families may work in more than one region and in different production areas depending on climate and time. Migration to the Black Sea region is carried out for the hazelnut harvest. During the hazelnut harvest, which can last from August to September 15, workers reside in Artvin, Rize, Trabzon, Giresun, Ordu, Samsun, Sinop, Zonguldak, Bartın, Sakarya, Kocaeli. Some of these workers additionally travel to Çukurova and other cotton-growing provinces in September-October for the cotton harvest.

According to the 2011 nationwide "Determination of the Needs of Seasonal Agricultural Workers and Their Families Survey", it was found that seasonal agricultural workers' needs mostly related to shelter such as toilets, bathrooms, hygiene, electricity/clean water, isolation, health services and childcare could not be adequately met. Seasonal agricultural workers work under many disadvantageous conditions.

There is a need for further studies on the physical and psychological effects of these harsh conditions in the open environment and in the summer season and the negative changes that may be caused by working as seasonal workers at a young age.

ELIGIBILITY:
Inclusion Criteria (For seasonal workers):

* Volunteering to participate in the study.
* To be between the ages of 18-34.
* Having worked as a seasonal worker in Giresun for at least 1 month during the hazelnut harvest period.

Inclusion Criteria (For controls):

* Volunteering to participate in the study.
* To be between the ages of 18-34.
* Not having worked in any agricultural work during the summer period.
* Living in the same socioeconomic environment as the group working as seasonal workers

Exclusion Criteria:

* Having visual, auditory, etc. communication problems that will prevent participation in the study.

Ages: 18 Years to 34 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Seasonal agricultural workers and not working control group in the same age and socioeconomic environment
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2024-09-01 (Actual); Primary Completion 2024-11-01 (Actual); Study Completion 2024-12-01 (Actual)

PRIMARY OUTCOMES:
McGill Melzack Questionnaire | Baseline
  Pain assessment (McGill Melzack Questionnaire) Participants' pain site, intensity and type will be assessed with the McGill-Melzack pain questionnaire. This questionnaire was first developed by Melzack and Katz in 1971. It consists of four parts. In part 1, there are two body pictures drawn from the front and back to mark the area or areas of the body affected by the patient's pain. The patient is asked to mark the location of the pain on the body diagram and indicate with the letter 'D' if the pain is deep and 'Y' if it is on the body surface. In the second part, the participant is asked to describe their pain. The participant marks the appropriate words from the appropriate group. A suitable word from each group can be marked or if it is not suitable, the group can be skipped altogether. In the third part, the relationship between pain and time is asked.
PhysioPrint Mobile Application | Baseline
  Posture assessment (PhysioPrint Mobile Application) The evaluation of the participants' posture will be performed with the PhysioPrint mobile application. The application has validity and reliability. The analysis is done by taking an image of the participant from the opposite side to assess posture disorders. The differences between the shoulder height levels, hip joint symmetry, and if there is hip joint symmetry, the differences between the kneecap alignments are determined angularly. The distance and angle of the foot and ankle joints to other anatomical regions can also be examined. After the analysis data is saved, the images will be deleted. In our study, this analysis will be used to compare the differences seen in seasonal workers with the non-working group.
Checklist Individual Strength Questionnaire | Baseline
  Fatigue assessment (Checklist Individual Strength Questionnaire) Fatigue will be assessed with the Fatigue Scale for both groups. The Fatigue Scale asks about fatigue in the two weeks prior to the assessment. It has 20 items, each item is scored on a seven-point Likert scale. A high score indicates high levels of subjective fatigue and concentration problems and low levels of motivation and physical activity. It has Turkish validity and reliability, and its internal consistency was reported to be high.

SECONDARY OUTCOMES:
Beck Depression Inventory | Baseline
  Mental State Assessment (Beck Depression Inventory) Participants' depression levels will be assessed with the Beck Depression Scale. It is a 21-item self-report questionnaire to assess the severity of depression in normal and psychiatric populations. It was developed by Beck et al. and revised in 1978. It is suitable for the assessment of the population aged 13 years and older. Each item is scored between 0-3 and the total score ranges between 0-63. A high score indicates a high level of depression.

CONTACTS AND LOCATIONS:
Locations (1):
- İstanbul BilgiUniversity, Istanbul, Beyoğlu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided